CLINICAL TRIAL: NCT06768814
Title: Overdose Recovery and Care Access (ORCA) Qualitative Stakeholder Interviews and County-level Data
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Caleb Banta-Green, Research Professor, School of Medicine, Psychiatry, University of Washington
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00019871; R33DA057600 (NIH)
Record Dates: First submitted 2025-01-06; First posted 2025-01-10 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Opioid Use Disorder; Opioid Use
Keywords: opioid overdose; opioid poisoning; harm-reduction; sub-acute stabilization
MeSH Terms: conditions — Opioid-Related Disorders; Opiate Overdose; Harm Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Other): The sub-acute stabilization center will combine: 1) post-overdose medical and social support, 2) the offer of starting medications for opioid use disorder, and 3) harm reduction services and supplies.
  Interventions: Behavioral: Sub-acute stabilization
- Comparison (No Intervention): Eligible Seattle EMS patients who opt not to go to the sub-acute stabilization center, and King County residents, outside of Seattle, who meet the same eligibility criteria.

INTERVENTIONS:
Behavioral: Sub-acute stabilization — The sub-acute stabilization center (SASC) is for people who have had or are at risk for having an opioid overdose and have an encounter with Seattle Fire Department emergency medical services (EMS) in Seattle, WA. Those transported to the SASC are the intervention participants and two comparison groups will be utilized: eligible Seattle EMS patients who opt not to go to the SASC and King County residents, outside of Seattle, who meet the same eligibility criteria. A comparative interrupted time series analysis is planned to study the main effectiveness outcomes. Seattle Fire EMS will assess, refer, and arrange transport participants to the SASC. The SASC will offer an array of services including post-overdose monitoring, utilization of buprenorphine and methadone for the treatment opioid use disorder and opioid withdrawal, linkage to ongoing care for OUD, and provision of harm reduction services and supplies. The length of stay in the SASC will be limited to less than 24 hours.
  Arms: Intervention

SUMMARY:
The study is a quasi-experimental investigation of a sub-acute stabilization center (SASC) for people who have had or are at risk for having an opioid overdose and have an encounter with Seattle Fire Department emergency medical services (EMS) in Seattle, WA. Those transported to the SASC are the intervention participants and two comparison groups will be utilized: eligible Seattle EMS patients who opt not to go to the SASC and King County residents, outside of Seattle, who meet the same eligibility criteria. A comparative interrupted time series analysis is planned to study the main effectiveness outcomes.

Seattle Fire EMS will assess, refer, and arrange transport for participants to the SASC. The SASC will offer an array of services including post-overdose monitoring, utilization of buprenorphine and methadone for the treatment opioid use disorder and opioid withdrawal, linkage to ongoing care for OUD, and provision of harm reduction services and supplies. The length of stay in the SASC will be limited to less than 24 hours. A continuous process improvement (CPI) approach will monitor and refine the intervention. Characterization of the interventions will be based upon analysis of service utilization patterns over time along with interviews and surveys with stakeholders.

DETAILED DESCRIPTION:
1. Clinical Intervention

   * We will be conducting a quasi-experimental study of a new sub-acute stabilization center (SASC) for those at high risk or who have had an opioid overdose to which Seattle Fire/EMS refer. All eligible people at risk or post OD who encounter Seattle Fire/EMS will potentially be offered the intervention, and those interested and transported will be considered study participants, there is no study assignment (anticipated n=5,495).
   * Comparison groups will be identified from secondary EMS records data for Seattle (anticipated n=7,223) and the remainder of King County, WA (anticipated n=11,550).
   * People 18 and older who EMS encounter who have had or are at high risk for any opioid overdose and meet clinical inclusion criteria.
   * SASC services will be provided by Downtown Emergency Service Center's Overdose Recovery and Care Access Centers:

     * 515 Third Avenue, Seattle, WA 98104
     * 517 Third Avenue, Seattle, WA 98104
     * 1600 South Lane Street Seattle, WA 98144
2. Implementation research interviews with professional stakeholders

   * We will be conducting repeated cross-sectional interviews with professional stakeholders about the implementation of the SASC and CPI activities.
   * Participants will be 18 or older and include people such as: CPI meeting attendees, EMS personnel, and SASC staff (n=60).
   * It is anticipated that stakeholder interviews will be conducted virtually via video conferencing with study team members.
3. Implementation research surveys with people with lived experience of drug use

   * We will be utilizing a combination of data sources. Initially in-person interview data from the 1R01DA059011-01 study (Van Draanen, PI) will be utilized for analyses.
   * Participants from the Van Draanen study will be 18 or older who have have survived a non-fatal opioid overdose and had an emergency medical service interaction or intervention (n=80).
   * If needed, we will also, subsequently conduct repeated cross-sectional surveys with people with lived experience of drug use about their experiences and perceptions of the SASC. Final procedures will be determined in collaboration with our community partner the Lived Expertise Advisory Board.

ELIGIBILITY:
Inclusion Criteria:

1. Verbally consents to transfer of care to SASC.
2. Awake and oriented to person and place, with no significant deficits in mental status or neurological function.
3. Age >=18
4. Patent airway and effective respirations with adequate oxygenation.
5. Stable heart rate and blood pressure, with no evidence of cardiac arrhythmias or other significant cardiovascular disfunction.
6. Vitals:

   * Heart rate: 45-130
   * Blood pressure: systolic 95-190, diastolic 50-120
   * Respiratory rate: 10-24
   * SpO2: >92 on room air or supplemental O2 via nasal cannula.
   * SpO2 <92% with supplemental O2 requires ED transfer.
   * EtCO2: <50
   * Temperature: 95.5-100.3 F
   * Blood glucose (if indicated): 60-300
7. No signs of head trauma:

   * Dizziness or loss of balance
   * Blurred vision or double vision
   * Sensitivity to light or noise
   * Seizures or convulsions
   * Weakness or numbness in the arms or legs
   * Persistent or worsening headache
   * CSF or blood leaking from the nose or ears
   * Unequal pupils or pupils that are slow to react to light.
8. No signs of other traumatic injury or medical needs requiring immediate treatment.
9. No signs of respiratory infection. Screen for COVID-19. See COVID-19 Screening protocol.

Exclusion Criteria:

- People under 18 and who do not meet SASC admission criteria will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40000 (Estimated)
Dates: Start 2024-12-15 (Actual); Primary Completion 2028-05-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Repeat opioid overdose | 1 year
  One of more opioid overdoses after enrollment
MOUD initiation | 1 year
  Starting opioid use disorder treatment with buprenorphine, methadone or naltrexone
MOUD retention | 1 year
  Having one or more additional doses prescribed, administered or dispensed of buprenorphine, methadone, or naltrexone
Emergency department utilization | 1 year
  Having one or more all-cause emergency department admission
EMS utilization | 1 year
  Having one or more emergency medical service encounters
Cost-effectiveness | 1 year
  Analysis from the perspective of a public sector payer of the per unit cost of reduced opioid overdoses attributable to the diversion program

OTHER OUTCOMES:
Service utilization patterns | 1 year
  Changes in the way services or opioid-related emergencies are provided and changes to cascade of care changes over time (descriptive).
Staff observations | 1 year
  How care opioid-related care is viewed by SASC staff members (descriptive).
Continuous process improvement (CPI) partner observations | 1 year
  How care opioid-related care is viewed by CPI partners and participants (descriptive).

CONTACTS AND LOCATIONS:
Overall Officials: Caleb Banta-Green, PhD, MPH, MSW, Principal Investigator — University of Washington
Locations (1):
- Downtown Emergency Service Center's Overdose Recovery and Care Access Centers, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No